CLINICAL TRIAL: NCT00579969
Title: Comparison of the Effects of Latanoprost and Timolol on Aqueous Humor Dynamics in Ocular Hypertensive Patients
Brief Title: Comparison of Latanoprost Vs. Timolol
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Study stopped and data not analyzed
Sponsor: University of Nebraska (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 0335-03-XX
Record Dates: First submitted 2007-12-18; First posted 2007-12-24 (Estimated); Last update posted 2023-12-21 (Actual); Status verified 2023-12

CONDITIONS: Glaucoma
MeSH Terms: conditions — Glaucoma | interventions — Latanoprost; Timolol

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Latanoprost Effects on Aqueous Humor Dynamics in Ocular Hypertensive Patients (Experimental): Evaluating the Effects of Latanoprost on Aqueous Humor Dynamics in Ocular Hypertensive Patients (prostaglandin analogue)
  Interventions: Drug: Latanoprost
- Timolol Effects on Aqueous Humor Dynamics in Ocular Hypertensive Patients (Experimental): Evaluating the Effects of Timolol on Aqueous Humor Dynamics in Ocular Hypertensive Patients (prostaglandin analogue)
  Interventions: Drug: Timolol

INTERVENTIONS:
Drug: Latanoprost — dosage form:eye drops, dosage: One drop in each eye twice a day
  Arms: Latanoprost Effects on Aqueous Humor Dynamics in Ocular Hypertensive Patients
Drug: Timolol — dosage form:eye drops, dosage: One drop in each eye twice a day
  Arms: Timolol Effects on Aqueous Humor Dynamics in Ocular Hypertensive Patients

SUMMARY:
The primary purpose of this study is to show, through a controlled masked clinical study of subjects with ocular hypertension (OHT), that latanoprost increases the low uveoscleral drainage of aqueous humor back to normal levels, and timolol maleate reduces the formation of aqueous humor below normal. Both of these mechanisms will effectively reduce intraocular pressure (IOP).

The secondary purpose is to assess the effects of both latanoprost and timolol maleate on the fluorophotometric outflow facility, and episcleral venous pressure and on all parameters over time.

DETAILED DESCRIPTION:
A recent publication by our laboratory has shown that patients with ocular hypertension (OHT) have reduced uveoscleral outflow and reduced trabecular outflow facility compared with healthy age-matched controls. These changes are the cause of the elevated intraocular pressure (IOP). Aqueous flow rate did not change in these patients. It is logical to assume that it would be more efficacious to treat OHT patients with drugs that reduce IOP by increasing uveoscleral outflow (which is abnormally low) than with drugs that reduce aqueous flow (which is normal in OHT).

The primary purpose of this study is to show, through a controlled masked clinical study of OHT patients, that latanoprost increases the low uveoscleral drainage of aqueous humor (Fu) back to normal levels, and timolol maleate reduces the formation of aqueous humor (Fa) below normal. Both of these mechanisms will effectively reduce IOP.

The secondary purpose is to assess the effects of both latanoprost and timolol maleate on the fluorophotometric outflow facility (Cflu), and episcleral venous pressure (Pev) and on all parameters over time.

Subjects eligible to participate will be at least 19 years of age and diagnosed with bilateral ocular hypertension or primary open angle glaucoma and have intraocular pressure between 20 and 35 mmHg in both eyes on Day 0. Subjects will be treated with either latanoprost or timolol for 6 weeks and then crossover and be treated similarly with the alternate drug for an additional 6 weeks. There will be a screening visit and a total of 6 study visits in which aqueous humor flow, uveoscleral outflow, and fluorophotometric outflow facility will be determined using an instrument called a fluorophotometer. The fluorophotometer scans the eye for fluorescein dye allowing the investigator to measure and calculate the above variables. There will be 7 scans taken during each study day and additionally IOP will be measured after the completion of each scan. An Exit exam will be performed at the time of exit to ensure the ocular health of the subject.

Subjects will be monitored for adverse events throughout the course of the study and subjects may discontinue from the study at any time for any reason, or may be discontinued if, in the opinion of the investigator, there is a risk to the subject.

ELIGIBILITY:
Inclusion Criteria:

* Minimum of nineteen (19) years of age.
* Diagnosed with bilateral ocular hypertension or primary open angle glaucoma for at least six months prior to screen visit.
* IOP of 20-35 mmHg in both eyes and not more than 5 mmHg difference between eyes at the Baseline 0800 ±1 hour IOP measurement.
* Willing and able to provide informed consent.
* Able to adhere to treatment/visit plan.

Exclusion Criteria:

Systemic Conditions:

* History of severe, unstable or uncontrolled cardiovascular, hepatic or renal disease.
* History of bronchial asthma or chronic obstructive pulmonary disease.
* Allergies to sulfa drugs.

Ocular Conditions:

* Chronic or recurrent severe ocular inflammatory disease.
* Ocular infection or inflammation within three (3) months of the study visit.
* Subjects currently treated with more than two ocular hypotensive medications.
* Subjects having previous exposure to: adrenergic antagonists, topical prostaglandin analogues (including latanoprost, unoprostone, travoprost and bimatoprost) within four (4) weeks of the baseline visit; adrenergic agonists within two (2) weeks of the baseline visit; and cholinergic agonists and carbonic anhydrase inhibitors within five (5) days of the baseline visit.
* History of any severe ocular pathology that would preclude the administration of a topical prostaglandin or beta-blocker.
* History of severe or serious hypersensitivity to topical or systemic prostaglandins or beta-blockers.
* Intraocular pressures less than 20 mmHg when off all ocular medications.
* Cornea thickness greater than 600 microns.

Women:

* Women of childbearing potential who are sexually active, or plan to become sexually active, and don't have a vasectomized partner, must agree to use at least one of the following acceptable contraceptive methods: condoms (male or female with or without a spermicidal agent, a diaphragm or cervical cap with spermicide, an intrauterine device (IUD) or hormonal-based contraception. Women of childbearing potential are defined as women who are not surgically sterile or not postmenopausal (at least 12 months without menstrual period).
* Nursing mothers.
* Pregnancy
* General
* Subjects less than nineteen (19) years of age.
* Therapy with another investigational agent within 30 days of Screening Visit.

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2003-12; Primary Completion 2008-10 (Actual); Study Completion 2008-10 (Actual)

PRIMARY OUTCOMES:
Comparison of Latanoprost and Timolol in lowering ocular pressure | 6 months
  Two drugs, Latanoprost and Timolol, will be compared in ocular hypertensive patients in their ability to lower ocular pressure at six months using a Goldmann applanation tonometer (GAT).

CONTACTS AND LOCATIONS:
Overall Officials: Carl B Camras, MD, Principal Investigator — UNMC Department of Ophthalmology
Locations (1):
- UNMC Department of Ophthalmolgy and Visual Sciences, Omaha, Nebraska, United States